CLINICAL TRIAL: NCT05314400
Title: A Prospective Study Evaluating Diagnostic Accuracy, Outcome, and Economic Impact of Abbreviated Gadoxetate-enhanced MRI of the Liver in Patients With Metastatic Colorectal Carcinoma
Brief Title: Gadoxetate Abbreviated MRI in Metastatic Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Harry Marshall, Assistant Professor of Radiology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 120191
Record Dates: First submitted 2022-03-17; First posted 2022-04-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: Colorectal Cancer; Liver Metastasis; Gadoxetate (Primovist / Eovist); Abbreviated MRI
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Full Protocol (Active Comparator): Routine Primovist MRI
  Interventions: Diagnostic Test: Full Gadoxetate-enhanced liver MRI
- Abbreviated Protocol (Experimental): Shortened Primovist MRI
  Interventions: Diagnostic Test: Shortened Gadoxetate-enhanced liver MRI

INTERVENTIONS:
Diagnostic Test: Full Gadoxetate-enhanced liver MRI — Standard pulse sequences
  Arms: Full Protocol
Diagnostic Test: Shortened Gadoxetate-enhanced liver MRI — Fewer pulse sequences
  Arms: Abbreviated Protocol

SUMMARY:
After a patient is diagnosed with colon cancer, they receive a CT of the chest, abdomen, and pelvis to see if the cancer has spread (metastasized) to other parts of the body. A common site for the cancer to spread to is the liver. If an abnormality is seen in the liver on CT, sometimes an MRI of the liver is required to determine a) whether it is cancer or not and b) whether there are small tumours in the liver that were not visible on CT.

During the MRI, the patient is injected with intravenous (IV) contrast. This makes liver lesions more conspicuous and also helps determine if they are cancerous or not. The most commonly used IV contrast agent is called Gadovist. However, there is another IV contrast agent called Primovist that is better at detecting liver metastases from colon cancer than Gadovist. This is very important information for surgeons, because if they considering cutting out (resecting) the liver tumours, they want to make sure they get them all.

Unfortunately, Primovist is used sparingly in Canadian hospitals because it is more expensive than Gadovist and the MRI takes longer. Some early small studies have suggested that it may be possible to shorten the Primovist MRI significantly (e.g. from 60 minutes to 15 minutes), making it economically feasible to offer Primovist to more patients. However, there have not been any large studies performed to confirm these findings.

The purpose of this study is to compare the accuracy of colon cancer liver metastasis detection between a regular, full-length Primovist MRI versus a shortened Primovist MRI protocol. The economic impact will also be assessed.

DETAILED DESCRIPTION:
BACKGROUND

Colorectal cancer (CRC) is the third most commonly diagnosed cancer in Canada and the second leading cause of death in both men, and women (1). In 2021, 24800 Canadians were diagnosed with CRC and 9,600 died from the disease (1). Over their lifetime, 1 in 18 Canadians will be diagnosed with CRC and 1 in 37 will die (1). Accurate staging is essential to improving outcomes, providing appropriate patient management, and improving the health care costs associated with caring for patients with CRC.

London Health Sciences Centre (LHSC) is a tertiary care referral centre for a catchment area of 2 million people in Southwestern Ontario. Annually, approximately 200 patients present to the London Regional Cancer Program with a diagnosis of colorectal cancer. Of these, about 100 patients will have potentially resectable colorectal liver metastasis (CRCLM).

Staging algorithms for CRC include contrast enhanced computed tomography (CECT) of the thorax/abdomen/pelvis, with MRI of the liver in some centres. The objective for performing imaging tests is to accurately determine the extent of local and distant disease to direct patient management. Accurate assessment of the hepatic disease burden is crucial for surgical planning since resection of liver metastases is a core component of CRCLM treatment (2). At LHSC, all patients are initially imaged with CECT of the thorax/abdomen/pelvis. MRI of the liver is reserved for patients that require further characterization of equivocal liver lesions detected on CT. When performed, liver MRI is often performed with extracellular agents such as gadobutrol (Gadovist), i.e. EC-MRI.

Hepatobiliary MRI contrast agents such as gadoxetic acid (aka gadoxetate, trade name Primovist in Canada), i.e. EOB-MRI, provide superior accuracy in detection of CRCLM compared to both CECT (3) and EC-MRI (4). Moreover, the use of EOB-MRI can alter management decisions and improve patient outcomes (3,5,6). It is also the modality of choice in CRCLM patients post-systemic therapy as per the 9th International Forum for Liver MRI Consensus Report (7).

Despite these data, hepatobiliary agents are being used sparingly in most Canadian hospitals, including at LHSC as a problem-solving tool. This is due to two factors: (a) the higher unit cost of gadoxetate compared to gadobutrol and iodine-based CT contrast agents, and (b) the increased MRI scan time required for EOB-MRI compared to EC-MRI or CECT. The increased scan time is a result of the need to acquire images in the "hepatobiliary (HPB) phase" for EOB-MRI, typically 20 minutes post-injection, a longer delay than is required for EC-MRI or CECT. These factors result in increased operational costs for EOB-MRI and opportunity costs from reduced magnet time for other MRI studies.

To address the increased scan time with EOB-MRI, some studies have retrospectively examined the potential role of abbreviated MRI protocols (aMRI) compared to a full protocol (fMRI) (8-11). The premise of EOB-aMRI protocols involves an injection of gadoxetate at the outset of the study, often outside the scanner room. During the 20 min waiting period prior to image acquisition in the HPB phase, an "abbreviated" set of sequences is acquired, usually including DWI/ADC and sometimes T2 weighted images. At the 20 min mark, the HPB phase images are acquired, and the study is complete. The aim of abbreviated protocols is to increase patient throughput without compromising diagnostic accuracy.

The initial results in this relatively nascent field are promising, showing high interobserver agreement and high diagnostic accuracy not significantly different from the full protocol. For example, Canellas et al reported both κ and area under the ROC curve (AUC) of greater than 0.9 for both aMRI and fMRI, with an estimated cost savings of 41% per scan (10). Ghorra et al found similar detection rates of about 86% for both aMRI and fMRI with slightly lower accuracy of the aMRI protocol of about 87% vs 93% for fMRI, but no consistent statistical trends were present (11).

However, existing studies in the literature have simulated an aMRI examination by using a subset of fMRI sequences; some sequences, including the dynamic post contrast sequences acquired before 20 min are removed retrospectively (8-11). Currently there are no published studies comparing fMRI with prospectively acquired aMRI. As retrospective studies may overestimate accuracy and cost savings, there is a need for higher quality, prospective evidence (7). Additionally, retrospective studies are unable to perform a formal economic analysis of costs related to the imaging procedure itself, and importantly downstream costs related to patient management.

RATIONALE

The primary aim of this study is to prospectively compare the diagnostic accuracy of aMRI compared to fMRI regarding CRCLM, using a composite reference standard. Our hypothesis is that aMRI is noninferior to fMRI in this regard, as measured by sensitivity, specificity, and the AUC. If this is the case, it may serve as evidence that EOB-MRI utilization can be increased even within resource constraints inherent to all Healthcare systems. The rationale for using a composite reference standard is that due to varying patient management strategies, the optimal reference standard (surgical pathology) is not always available, and therefore alternative methods must be considered. The rationale for using fMRI as the control group is that this protocol is the current standard of care for EOB-MRI.

A secondary aim is to quantify the economic impact of aMRI vs fMRI both in terms of imaging costs and downstream patient management costs. Our hypothesis is that aMRI will not cost more than fMRI on a per patient basis (i.e. noninferiority). If this is the case, higher patient throughput can be achieved at no increased economic expense.

A second secondary aim is to evaluate patient outcomes (overall survival, cancer-specific survival, and hepatic recurrence / progression free survival) at 1-year post-baseline EOB-MRI, using clinical data and the 1-year follow-up CECT. Our hypothesis is that aMRI will be noninferior to fMRI, indicating that there is no adverse effect on patient outcomes from the using an abbreviated protocol.

The third secondary aim is to retrospectively compare the diagnostic accuracy of fMRI to a simulated aMRI created from a subset of fMRI pulse sequences. Our hypothesis is that the simulated aMRI will be noninferior to fMRI. This constitutes a 3-factor multireader multicase design, analogous to multiple prior investigations (3,4), enabling direct comparison of our study and adding to the body of literature on the subject.

The final study aim is to compare the diagnostic accuracy and interobserver agreement on aMRI and fMRI. Our hypothesis is that there will be no significant difference for diagnostic accuracy. We expect interobserver agreement to be moderate to high.

The rationale for choosing a study cohort comprised of patients with CRCLM is: 1) this is a large patient population / common patient presentation, and 2) EOB-MRI has been shown to provide added value for staging CRCLM but is likely underutilized in Canada, as detailed above.

The rationale for choosing a 1-year follow-up period is that about 30% to 50% of CRCLM will recur or progress within this interval (12,13), enabling a compromise between capturing a significant portion of adverse patient outcomes while minimizing loss to follow-up and unnecessarily prolonging the study, as this is not the primary objective.

STUDY DESIGN

This is a prospective, block randomized, allocation concealed, unblinded, multireader study with case-nested-within-test split-plot design.

The baseline abbreviated or full Primovist MRI will be acquired between day 2 and 14 and a follow-up contrast enhanced CT abdomen pelvis will be performed 1 year from baseline. A combination of histopathology, biological behavior, and imaging findings applied in a hierarchical manner will determine the reference standard for each focal hepatic lesion, i.e. metastasis or not. Sample size is 200 subjects, with equal distribution of 100 per arm.

Statistical analysis of the primary endpoint will be conducted via the updated Obuchowski-Rockette (OR) method (14).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Diagnosis of colorectal cancer, biopsy proven
* Prior imaging showing liver lesions that may be metastases
* Provision of signed and dated informed consent form
* Willingness to comply with study procedures and availability for the duration of the study
* Able to tolerate MRI required by protocol

Exclusion Criteria:

* Presence of implanted medical device or metallic object that is MR incompatible
* Baseline eGFR of < 30 mL/min/1.73 m2
* Severe claustrophobia not relieved by oral anxiolytics
* Documented severe allergic-like reaction gadolinium-based contrast agent
* Weight greater than allowable on MRI table
* Pregnancy
* Diffuse liver metastases, i.e. definitively unresectable
* Severe liver dysfunction, ALBI grade 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of abbreviated versus full MRI protocol | 2 years
  Sensitivity, specificity, area under ROC curve

SECONDARY OUTCOMES:
Cost of abbreviated versus full MRI protocol | 3 years
  Sum of the following dollar amounts: technical MRI fees + professional MRI fees + MRI time (cost per hour defined by local institution * number hours used)
Overall survival at 1 year post abbreviated versus full MRI protocol | 3 years
  Proportion of patients alive at 1 year (dimensionless)
Cancer specific survival at 1 year post abbreviated versus full MRI protocol | 3 years
  1 - proportion of patients who died of colorectal cancer or its complications (dimensionless)
Progression free survival at 1 year post abbreviated versus full MRI protocol | 3 years
  1 - proportion of patients with evidence of recurrent or progressive hepatic disease at 1 year (dimensionless)
Diagnostic accuracy of simulated abbreviated versus full MRI protocol | 2 years
  Sensitivity, specificity, area under ROC curve
Inter-reader agreement for all modalities | 2 years
  Sensitivity, specificity, area under ROC curve, and kappa coefficient

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare, London, Ontario
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Cancer Statistics Advisory Committee in collaboration with the Canadian Cancer Society, Statistics Canada and the Public Health Agency of Canada. (2021).
- [Background] Yamamoto M, Yoshida M, Furuse J, Sano K, Ohtsuka M, Yamashita S, Beppu T, Iwashita Y, Wada K, Nakajima TE, Sakamoto K, Hayano K, Mori Y, Asai K, Matsuyama R, Hirashita T, Hibi T, Sakai N, Tabata T, Kawakami H, Takeda H, Mizukami T, Ozaka M, Ueno M, Naito Y, Okano N, Ueno T, Hijioka S, Shikata S, Ukai T, Strasberg S, Sarr MG, Jagannath P, Hwang TL, Han HS, Yoon YS, Wang HJ, Luo SC, Adam R, Gimenez M, Scatton O, Oh DY, Takada T. Clinical practice guidelines for the management of liver metastases from extrahepatic primary cancers 2021. J Hepatobiliary Pancreat Sci. 2021 Jan;28(1):1-25. doi: 10.1002/jhbp.868. Epub 2020 Dec 12. PMID 33200538
- [Background] Vreugdenburg TD, Ma N, Duncan JK, Riitano D, Cameron AL, Maddern GJ. Comparative diagnostic accuracy of hepatocyte-specific gadoxetic acid (Gd-EOB-DTPA) enhanced MR imaging and contrast enhanced CT for the detection of liver metastases: a systematic review and meta-analysis. Int J Colorectal Dis. 2016 Nov;31(11):1739-1749. doi: 10.1007/s00384-016-2664-9. Epub 2016 Sep 29. PMID 27682648
- [Background] Choi SH, Kim SY, Park SH, Kim KW, Lee JY, Lee SS, Lee MG. Diagnostic performance of CT, gadoxetate disodium-enhanced MRI, and PET/CT for the diagnosis of colorectal liver metastasis: Systematic review and meta-analysis. J Magn Reson Imaging. 2018 May;47(5):1237-1250. doi: 10.1002/jmri.25852. Epub 2017 Sep 13. PMID 28901685
- [Background] Kim C, Kim SY, Kim MJ, Yoon YS, Kim CW, Lee JH, Kim KP, Lee SS, Park SH, Lee MG. Clinical impact of preoperative liver MRI in the evaluation of synchronous liver metastasis of colon cancer. Eur Radiol. 2018 Oct;28(10):4234-4242. doi: 10.1007/s00330-018-5422-2. Epub 2018 Apr 24. PMID 29691635
- [Background] Jhaveri KS, Fischer SE, Hosseini-Nik H, Sreeharsha B, Menezes RJ, Gallinger S, Moulton CE. Prospective comparison of gadoxetic acid-enhanced liver MRI and contrast-enhanced CT with histopathological correlation for preoperative detection of colorectal liver metastases following chemotherapy and potential impact on surgical plan. HPB (Oxford). 2017 Nov;19(11):992-1000. doi: 10.1016/j.hpb.2017.06.014. Epub 2017 Jul 29. PMID 28760631
- [Background] Koh DM, Ba-Ssalamah A, Brancatelli G, Fananapazir G, Fiel MI, Goshima S, Ju SH, Kartalis N, Kudo M, Lee JM, Murakami T, Seidensticker M, Sirlin CB, Tan CH, Wang J, Yoon JH, Zeng M, Zhou J, Taouli B. Consensus report from the 9th International Forum for Liver Magnetic Resonance Imaging: applications of gadoxetic acid-enhanced imaging. Eur Radiol. 2021 Aug;31(8):5615-5628. doi: 10.1007/s00330-020-07637-4. Epub 2021 Feb 1. PMID 33523304
- [Background] Kim JW, Lee CH, Park YS, Lee J, Kim KA. Abbreviated Gadoxetic Acid-enhanced MRI with Second-Shot Arterial Phase Imaging for Liver Metastasis Evaluation. Radiol Imaging Cancer. 2019 Sep 27;1(1):e190006. doi: 10.1148/rycan.2019190006. eCollection 2019 Sep. PMID 33778670
- [Background] Granata V, Fusco R, Avallone A, Cassata A, Palaia R, Delrio P, Grassi R, Tatangelo F, Grazzini G, Izzo F, Petrillo A. Abbreviated MRI protocol for colorectal liver metastases: How the radiologist could work in pre surgical setting. PLoS One. 2020 Nov 19;15(11):e0241431. doi: 10.1371/journal.pone.0241431. eCollection 2020. PMID 33211702
- [Background] Canellas R, Patel MJ, Agarwal S, Sahani DV. Lesion detection performance of an abbreviated gadoxetic acid-enhanced MRI protocol for colorectal liver metastasis surveillance. Eur Radiol. 2019 Nov;29(11):5852-5860. doi: 10.1007/s00330-019-06113-y. Epub 2019 Mar 19. PMID 30888485
- [Background] Ghorra C, Pommier R, Piveteau A, Rubbia-Brandt L, Vilgrain V, Terraz S, Ronot M. The diagnostic performance of a simulated "short" gadoxetic acid-enhanced MRI protocol is similar to that of a conventional protocol for the detection of colorectal liver metastases. Eur Radiol. 2021 Apr;31(4):2451-2460. doi: 10.1007/s00330-020-07344-0. Epub 2020 Oct 6. PMID 33025173
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Mauer M, Tanis E, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative FOLFOX4 chemotherapy and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC 40983): long-term results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1208-15. doi: 10.1016/S1470-2045(13)70447-9. Epub 2013 Oct 11. PMID 24120480
- [Background] Yan TD, Sim J, Black D, Niu R, Morris DL. Systematic review on safety and efficacy of repeat hepatectomy for recurrent liver metastases from colorectal carcinoma. Ann Surg Oncol. 2007 Jul;14(7):2069-77. doi: 10.1245/s10434-007-9388-6. Epub 2007 Apr 14. PMID 17440785
- [Background] Obuchowski NA, Beiden SV, Berbaum KS, Hillis SL, Ishwaran H, Song HH, Wagner RF. Multireader, multicase receiver operating characteristic analysis: an empirical comparison of five methods. Acad Radiol. 2004 Sep;11(9):980-95. doi: 10.1016/j.acra.2004.04.014. PMID 15350579
- See also: Link to citation 1 (Canadian Cancer Statistics) — https://cdn.cancer.ca/-/media/files/research/cancer-statistics/2021-statistics/2021-pdf-en-final.pdf?rev=2b9d2be7a2d34c1dab6a01c6b0a6a32d&hash=01DE85401DBF0217F8B64F2B7DF43986